CLINICAL TRIAL: NCT05184829
Title: A Single-center Study on the Effect of Systemic/Selective Lymph Node Dissection on the Prognosis of Ground Glass Nodules Smaller Than 3cm and With Components With Consolidation/Tumor Ratio Between 0.5-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B2021
Record Dates: First submitted 2021-12-15; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Progression; Postoperative Recovery
MeSH Terms: conditions — Disease Progression

STUDY DESIGN:
Intervention Model Description: systemic or selective lymph node dissection group
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- systemic lymph node dissection group (Active Comparator): systemic lymph node dissection group
  Interventions: Other: Systemic Lymph Node Dissection
- selective lymph node dissection (Experimental): selective lymph node dissection
  Interventions: Other: selective lymph node dissection

INTERVENTIONS:
Other: selective lymph node dissection — selective lymph node dissection
  Arms: selective lymph node dissection
Other: Systemic Lymph Node Dissection — Systemic Lymph Node Dissection
  Arms: systemic lymph node dissection group

SUMMARY:
A single-center study on the effect of systemic/selective lymph node dissection on the prognosis of ground glass nodules smaller than 3cm and with components with consolidation/tumor ratio between 0.5-1

DETAILED DESCRIPTION:
A single-center study on the effect of systemic/selective lymph node dissection on the prognosis of ground glass nodules smaller than 3cm and with components with consolidation/tumor ratio between 0.5-1

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in the study must meet all of the following conditions:

* 1.Aged between 25 and 75 years;
* 2. GGO is diagnosed by thin-section lung CT (thickness <1.5mm) within one month before surgery;
* 3. The maximum diameter of the GGO is smaller than 3cm;
* 4. The solid component in GGO between 50%-100%;
* 5. Preoperative examination showed that the patient could tolerate lobectomy;
* 6. The patient is able to understand and comply with the study and has provided written informed consent.

Exclusion Criteria:

Patients meeting any of the following criteria are not eligible for this trial:

* 1. Patients with a history of lung surgery;
* 2. Postoperative pathology showed non-primary lung cancer;
* 3. The scope of surgical resection is larger than one lung lobe;
* 4. Patients with a history of other tumors;
* 5. Patients with severe complications (coronary heart disease, valvular heart disease, end-stage renal disease, severe liver cirrhosis);
* 6. Unable to cooperate with the researchers because of dementia or cognitive decline
* 7. Other situations that are not in conformity with the standards and requirements of this trial.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From enrollment to 36 months after surgery

SECONDARY OUTCOMES:
Complications | 1-2 Weeks after enrollment (after Surgery)
  The degrees of cough